CLINICAL TRIAL: NCT04919668
Title: The Effect of Gamification in an Online Grocery Store Experiment on Food Selection: a Randomized Controlled Trial
Brief Title: Effect of Gamification in an Online Grocery Store.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Duke University (Other); Wal-Mart Foundation (Unknown)
Responsible Party: Principal Investigator, Sean Cash, Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00001028
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Food Selection; Food Preferences; Behavior, Eating
Keywords: Gamification
MeSH Terms: conditions — Food Preferences; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low budget; no game (Sham Comparator): Participants will be asked to shop for 12 list items in the simulated grocery store without game elements (crowns and scoreboards) displayed. They will be given a low budget of $30.
  Interventions: Behavioral: Simulated grocery shopping exercise
- High budget; no game (Active Comparator): Participants will be asked to shop for 12 list items in the simulated grocery store without game elements (crowns and scoreboards) displayed. They will be given a high budget of $50.
  Interventions: Behavioral: Simulated grocery shopping exercise
- Low budget; game (Active Comparator): Participants will be asked to shop for 12 list items in the simulated grocery store with game elements (crowns and scoreboards) displayed. They will be given a low budget of $30.
  Interventions: Behavioral: Simulated grocery shopping exercise
- High budget; game (Active Comparator): Participants will be asked to shop for 12 list items in the simulated grocery store with game elements (crowns and scoreboards) displayed. They will be given a high budget of $50.
  Interventions: Behavioral: Simulated grocery shopping exercise

INTERVENTIONS:
Behavioral: Simulated grocery shopping exercise — Participants will click a link and simulate an online grocery shopping experience by selecting items for 12 grocery categories.

SUMMARY:
The overall objective of this research is to evaluate the impact of gamification on the diet quality of food choices made by American adults in an online grocery shopping experiment. Participants will shop for 12 food items from a grocery shopping list determined by the research team in a simulated online grocery store designed for this experiment. Each product has a nutritional quality score based on the Guiding Stars algorithm. The experiment tests the gamification of the nutritional quality score. Participants exposed to gamification see one to five crowns illustrating the nutritional quality of the food and a scoreboard indicating the total number of crowns from foods in the participant's shopping basket. Participants will be assigned to experimental conditions of gamification (game or no game) and a fictitious budget ($30 or $50). The investigators will test if the game and the budget affect the dietary quality of their final shopping baskets. The experiment is a 2x2 experimental design. The investigators hypothesize that the presence of gamification will change the dietary quality of participants' final shopping baskets. The investigators hypothesize that a higher budget will change the dietary quality of the final shopping basket. The investigators also hypothesize that the game and higher budget together will change the dietary quality of the final shopping basket.

DETAILED DESCRIPTION:
Participants will be assigned to one of four experimental conditions:

1. Game=No and Budget = $30
2. Game=No and Budget = $50
3. Game=Yes and Budget = $30
4. Game=Yes and Budget = $50.

Variables:

1. Game: Indicates exposure to the game (dummy variable)
2. Budget: Indicates exposure low ($30) or high ($50) budget constraint (dummy variable).
3. Total number of crowns: sum of the number of crowns associated with the 12 items included in participants' final shopping baskets (a continuous variable that ranges from 12 to 60).
4. Number of crowns: number of crowns associated with each of the 12 items included in participants' final shopping baskets separately (a continuous variable that ranges from 1 to 5).

ELIGIBILITY:
The investigators will exclude from the analysis:

1. Participants who had more than or less than 12 items in their final shopping cart.
2. Participants who had four or more items from the same food subcategory in the final shopping basket.
3. Participants who spent more than 120% of the budget assigned to them.
4. Aged < 18 years
5. Do not have access to a personal computer, laptop, tablet, or mobile phone.
6. Participants who were not in the US when participating in the study.

Inclusion criteria:

1. Participants who had 12 items in their final shopping cart.
2. Participants who had less than four items from the same food subcategory in their final shopping basket.
3. Participants who spent 120% or less of the budget assigned to them.
4. Aged 18 or older
5. Have access to a personal computer, laptop, tablet, or mobile phone.
6. Participants who were in the US when participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1185 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Total number of crowns | One hour
  Sum of number of crowns of foods included in the final shopping basket for each participant

SECONDARY OUTCOMES:
Number of crowns | One hour
  Number of crowns for foods included in final shopping basket for each list item separately

OTHER OUTCOMES:
Total Guiding Stars points | One hour
  Sum of Guiding Stars points from foods included in the final shopping basket for each participant
Guiding Stars points | One hour
  Number of Guiding Stars points for foods included in final shopping basket for each list item separately

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data collected in this experiment will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication, or as required by a condition of awards and agreements supporting the research.
Access Criteria: Data will be available upon reasonable request. Proposals may be submitted up to 36 months of article publication. After 36 months, the data will be available at Tufts University data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Derived] Braga BC, Cash SB, Sarson K, Chang R, Mosca A, Wilson NLW. The gamification of nutrition labels to encourage healthier food selection in online grocery shopping: A randomized controlled trial. Appetite. 2023 Sep 1;188:106610. doi: 10.1016/j.appet.2023.106610. Epub 2023 Jun 2. PMID 37269883